CLINICAL TRIAL: NCT05065424
Title: Use of Premedication for Less Invasive Surfactant Administration: A Randomized Control Trial
Brief Title: Premedication for Less Invasive Surfactant Administration Study (PRELISA)
Acronym: PRELISA
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: Adverse event
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Principal Investigator, Venkat Kakkilaya, Principal Investigator, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STU-2021-0380
Record Dates: First submitted 2021-09-13; First posted 2021-10-04 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Respiratory Distress Syndrome, Newborn
Keywords: Premedication for Less Invasive Surfactant Administration; Fentanyl and Atropine for Less Invasive Surfactant Administration; Cerebral Near Infrared Spectroscopy monitoring in neonates; Premedication for LISA; Fentanyl and Atropine for LISA; Cerebral NIRS monitoring in neonates
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn | interventions — Atropine; Fentanyl

STUDY DESIGN:
Intervention Model Description: Quadruple Blinded
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IV Atropine and Fentanyl Premedication Arm (Experimental): Participants will receive premedication regimen of 20 micrograms/kilogram intravenous atropine and 0.5 micrograms/kilogram intravenous fentanyl prior to performance of LISA.
  Interventions: Drug: IV Atropine and Fentanyl Premedication Arm
- IV Normal Saline Placebo Arm (Placebo Comparator): Participants will receive two intravenous Normal Saline infusions in quantities equivalent to the calculated volumes of atropine and fentanyl for participant's weight prior to performance of LISA.
  Interventions: Drug: IV Normal Saline Placebo Arm

INTERVENTIONS:
Drug: IV Atropine and Fentanyl Premedication Arm — Prior to the LISA procedure, the blinded bedside nurse will infuse IV Atropine, labelled as "Atropine/Placebo," over 1 minute, followed by IV fentanyl, labelled as "Fentanyl/Placebo," over 20 minutes in the presence of blinded respiratory therapist and primary team provider.
  After medication infusion, a primary team member will perform Less Invasive Surfactant Administration procedure. Infant vital signs, cerebral Near Infrared Spectroscopy values, pain scores will be monitored and recorded during and for 12 hours after the procedure. Level of respiratory support, oxygen requirement and subsequent need for intubation for 24 hours after the procedure will be obtained from the electronic medical record.
  Other Names: IV Atropine sulfate and IV Fentanyl citrate
  Arms: IV Atropine and Fentanyl Premedication Arm
Drug: IV Normal Saline Placebo Arm — Prior to the Less Invasive Surfactant Administration procedure, the blinded bedside nurse will infuse IV Normal Saline, labelled as "Atropine/Placebo," over 1 minute, followed by a second infusion of IV Normal Saline, labelled as "Fentanyl/Placebo," over 20 minutes in the presence of blinded respiratory therapist and primary team provider.
  After Normal Saline infusion, primary team member will perform Less Invasive Surfactant Administration procedure. Infant vital signs, cerebral Near Infrared Spectroscopy values, pain scores will be monitored and recorded during and for 12 hours after the procedure. Level of respiratory support, oxygen requirement and subsequent need for intubation for 24 hours after the procedure will be obtained from the electronic medical record.
  Arms: IV Normal Saline Placebo Arm

SUMMARY:
The purpose of this study is to conduct a double blinded randomized control trial to determine the safety and efficacy of using IV fentanyl and atropine prior to Less Invasive Surfactant Administration (LISA) procedure in preterm infants with Respiratory Distress Syndrome compared to the local standard of care to perform this procedure without any premedication.

Hypothesis: In infants greater than or equal to 29 weeks gestational age requiring the Less Invasive Surfactant Administration procedure, premedication with a combination of IV atropine and IV fentanyl will be associated with fewer combined bradycardia events, defined as heartrate less than 100 beats per minute for longer than 10 seconds, and hypoxemia events, defined as saturations less than or equal to 80% for longer than 30 seconds, during the procedure compared with placebo.

Specific Aims:

* To determine if infants ≥29 week GA receiving IV fentanyl and atropine prior to LISA will have a decrease in hypoxemia and bradycardia events during the procedure compared to infants receiving placebo
* To determine if infants ≥29 week GA receiving premedication prior to Less Invasive Surfactant Administration will have higher procedure first attempt success rate compared with infants receiving placebo
* To determine the effect of premedication on cerebral oxygenation compared to placebo during and for 12 hours after Less Invasive Surfactant Administration in infants ≥29 week GA using cerebral Near Infrared Spectroscopy.
* To determine the effect of premedication prior to Less Invasive Surfactant Administration on the need for mechanical ventilation during ≤72 hours of life in preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* Infants ≥29 weeks gestational age initiated on CPAP in the delivery room or upon admission who require ≥0.25 FiO2.

Exclusion Criteria:

* Infants requiring intubation prior to surfactant therapy
* Infants with known severe congenital anomalies (including complex congenital heart disease, airway, and central nervous system anomalies)
* Infants born to mothers with known opioid addiction or in a methadone treatment program
* Maternal COVID19 infection (RT-PCR positive) within two weeks prior to delivery

Ages: 0 Hours to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of bradycardia and hypoxemia events during LISA procedure | Time of medication infusion to completion of LISA procedure
  * Bradycardia events will be defined as heartrate <100 beats per minute for >10 seconds. Heartrate will be obtained from the participant's heartrate monitor.
  * Hypoxemia events will be defined as participant saturation (SpO2) =<80% for >30 seconds. SpO2 will be obtained from the participant's pulse oximeter monitor.
  * Events will be recorded by the respiratory therapist and/ or bedside nurse present during the procedure

SECONDARY OUTCOMES:
Percent of time spent with cerebral Near Infrared Spectroscopy (NIRS) values <55% | From time of start of LISA procedure to 12 hours after procedure
  Cerebral NIRS is a method of noninvasively monitoring cerebral oxygenation. The probes detect a value every 6 seconds and display onto the monitor. Scores between 55-80% are considered within the normal range. Scores less than 55% are considered suboptimal cerebral oxygenation.
  * Percent of time spent with low NIRS values <55% during the 12 hour observation period will be calculated
Procedure first attempt success rate | At time of LISA procedure
  * Procedure attempt is defined as introduction of laryngoscope blade into the mouth.
  * Procedure success is defined by ability to insert catheter and administer surfactant, without surfactant aspirated from the stomach after administration.
  * Rate will be calculated as a percent of participants in each arm.
Intubation rate | Within 24 hours after LISA procedure
  * Rate will be calculated as a percent of participants in each group.
  * Participants need for and timing of intubation will be obtained from electronic medical record.
Mean number of attempts required | At time of LISA procedure
  Procedure attempt defined as introduction of laryngoscope blade into the mouth
Mean duration of bradycardia and hypoxemia events | Time of medication infusion to completion of LISA procedure
  * Bradycardia events will be defined as heartrate <100 beats per minute for >10 seconds. Heartrate will be obtained from the participant's heartrate monitor.
  * Hypoxemia events will be defined as participant saturation (SpO2) =<80% for >30 seconds. SpO2 will be obtained from the participant's pulse oximeter monitor.
  * Duration of events in seconds will be recorded by the respiratory therapist and/ or bedside nurse present during the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Venkatakrishna Kakkilaya, MD, Study Director — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Health and Hospital System, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdel-Latif ME, Davis PG, Wheeler KI, De Paoli AG, Dargaville PA. Surfactant therapy via thin catheter in preterm infants with or at risk of respiratory distress syndrome. Cochrane Database Syst Rev. 2021 May 10;5(5):CD011672. doi: 10.1002/14651858.CD011672.pub2. PMID 33970483
- [Background] Anand KJ; International Evidence-Based Group for Neonatal Pain. Consensus statement for the prevention and management of pain in the newborn. Arch Pediatr Adolesc Med. 2001 Feb;155(2):173-80. doi: 10.1001/archpedi.155.2.173. PMID 11177093
- [Background] Boggini T, Pozzoli S, Schiavolin P, Erario R, Mosca F, Brambilla P, Fumagalli M. Cumulative procedural pain and brain development in very preterm infants: A systematic review of clinical and preclinical studies. Neurosci Biobehav Rev. 2021 Apr;123:320-336. doi: 10.1016/j.neubiorev.2020.12.016. Epub 2020 Dec 20. PMID 33359095
- [Background] Bourgoin L, Caeymaex L, Decobert F, Jung C, Danan C, Durrmeyer X. Administering atropine and ketamine before less invasive surfactant administration resulted in low pain scores in a prospective study of premature neonates. Acta Paediatr. 2018 Jul;107(7):1184-1190. doi: 10.1111/apa.14317. Epub 2018 Apr 16. PMID 29532502
- [Background] Brummelte S, Grunau RE, Chau V, Poskitt KJ, Brant R, Vinall J, Gover A, Synnes AR, Miller SP. Procedural pain and brain development in premature newborns. Ann Neurol. 2012 Mar;71(3):385-96. doi: 10.1002/ana.22267. Epub 2012 Feb 28. PMID 22374882
- [Background] Committee on Fetus and Newborn; American Academy of Pediatrics. Respiratory support in preterm infants at birth. Pediatrics. 2014 Jan;133(1):171-4. doi: 10.1542/peds.2013-3442. Epub 2013 Dec 30. PMID 24379228
- [Background] Chevallier M, Durrmeyer X, Ego A, Debillon T; PROLISA Study Group. Propofol versus placebo (with rescue with ketamine) before less invasive surfactant administration: study protocol for a multicenter, double-blind, placebo controlled trial (PROLISA). BMC Pediatr. 2020 May 8;20(1):199. doi: 10.1186/s12887-020-02112-x. PMID 32384914
- [Background] Dekker J, Lopriore E, van Zanten HA, Tan RNGB, Hooper SB, Te Pas AB. Sedation during minimal invasive surfactant therapy: a randomised controlled trial. Arch Dis Child Fetal Neonatal Ed. 2019 Jul;104(4):F378-F383. doi: 10.1136/archdischild-2018-315015. Epub 2018 Aug 1. PMID 30068669
- [Background] Descamps CS, Chevallier M, Ego A, Pin I, Epiard C, Debillon T. Propofol for sedation during less invasive surfactant administration in preterm infants. Arch Dis Child Fetal Neonatal Ed. 2017 Sep;102(5):F465. doi: 10.1136/archdischild-2017-312791. Epub 2017 May 8. No abstract available. PMID 28483817
- [Background] Duerden EG, Grunau RE, Guo T, Foong J, Pearson A, Au-Young S, Lavoie R, Chakravarty MM, Chau V, Synnes A, Miller SP. Early Procedural Pain Is Associated with Regionally-Specific Alterations in Thalamic Development in Preterm Neonates. J Neurosci. 2018 Jan 24;38(4):878-886. doi: 10.1523/JNEUROSCI.0867-17.2017. Epub 2017 Dec 18. PMID 29255007
- [Background] Hyttel-Sorensen S, Pellicer A, Alderliesten T, Austin T, van Bel F, Benders M, Claris O, Dempsey E, Franz AR, Fumagalli M, Gluud C, Grevstad B, Hagmann C, Lemmers P, van Oeveren W, Pichler G, Plomgaard AM, Riera J, Sanchez L, Winkel P, Wolf M, Greisen G. Cerebral near infrared spectroscopy oximetry in extremely preterm infants: phase II randomised clinical trial. BMJ. 2015 Jan 5;350:g7635. doi: 10.1136/bmj.g7635. PMID 25569128
- [Background] Johnston L, Kwon SH. Moving from controversy to consensus: premedication for neonatal intubation. J Perinatol. 2018 Jun;38(6):611-613. doi: 10.1038/s41372-018-0115-x. Epub 2018 Jun 22. No abstract available. PMID 29930326
- [Background] Klotz D, Porcaro U, Fleck T, Fuchs H. European perspective on less invasive surfactant administration-a survey. Eur J Pediatr. 2017 Feb;176(2):147-154. doi: 10.1007/s00431-016-2812-9. Epub 2016 Dec 9. PMID 27942865
- [Background] Kumar P, Denson SE, Mancuso TJ; Committee on Fetus and Newborn, Section on Anesthesiology and Pain Medicine. Premedication for nonemergency endotracheal intubation in the neonate. Pediatrics. 2010 Mar;125(3):608-15. doi: 10.1542/peds.2009-2863. Epub 2010 Feb 22. PMID 20176672
- [Background] Kurepa D, Perveen S, Lipener Y, Kakkilaya V. The use of less invasive surfactant administration (LISA) in the United States with review of the literature. J Perinatol. 2019 Mar;39(3):426-432. doi: 10.1038/s41372-018-0302-9. Epub 2019 Jan 11. PMID 30635595
- [Background] Maheshwari R, Tracy M, Badawi N, Hinder M. Neonatal endotracheal intubation: How to make it more baby friendly. J Paediatr Child Health. 2016 May;52(5):480-6. doi: 10.1111/jpc.13192. PMID 27329901
- [Background] McPherson C, Grunau RE. Neonatal pain control and neurologic effects of anesthetics and sedatives in preterm infants. Clin Perinatol. 2014 Mar;41(1):209-27. doi: 10.1016/j.clp.2013.10.002. Epub 2013 Dec 17. PMID 24524456
- [Background] Rigo V, Lefebvre C, Broux I. Surfactant instillation in spontaneously breathing preterm infants: a systematic review and meta-analysis. Eur J Pediatr. 2016 Dec;175(12):1933-1942. doi: 10.1007/s00431-016-2789-4. Epub 2016 Sep 27. PMID 27678511
- [Background] Stow PJ, McLeod ME, Burrows FA, Creighton RE. Anterior fontanelle pressure responses to tracheal intubation in the awake and anaesthetized infant. Br J Anaesth. 1988 Feb;60(2):167-70. doi: 10.1093/bja/60.2.167. PMID 3345277
- [Background] Subramaniam P, Ho JJ, Davis PG. Prophylactic nasal continuous positive airway pressure for preventing morbidity and mortality in very preterm infants. Cochrane Database Syst Rev. 2016 Jun 14;(6):CD001243. doi: 10.1002/14651858.CD001243.pub3. PMID 27315509
- [Background] Sweet DG, Carnielli V, Greisen G, Hallman M, Ozek E, Te Pas A, Plavka R, Roehr CC, Saugstad OD, Simeoni U, Speer CP, Vento M, Visser GHA, Halliday HL. European Consensus Guidelines on the Management of Respiratory Distress Syndrome - 2019 Update. Neonatology. 2019;115(4):432-450. doi: 10.1159/000499361. Epub 2019 Apr 11. PMID 30974433